CLINICAL TRIAL: NCT02204098
Title: A Phase 1B Clinical Trial to Evaluate the Safety and Immune Response to a Mammaglobin-A DNA Vaccine in ER+, HER2- Breast Cancer Patients Undergoing Neoadjuvant Endocrine Therapy or Chemotherapy
Brief Title: Safety and Immune Response to a Mammaglobin-A DNA Vaccine In Breast Cancer Patients Undergoing Neoadjuvant Endocrine Therapy
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Rising Tide Foundation (Other); United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201407100; W81XWH-15-1-0101 (Other Grant/Funding Number: United States Department of Defense)
Record Dates: First submitted 2014-07-23; First posted 2014-07-30 (Estimated); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Breast Cancer; Breast Carcinoma; Malignant Neoplasm of Breast
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort 1:Neoadjuvant endocrine therapy alone (Active Comparator): * Will be treated with standard of care adjuvant endocrine therapy as determined by their treating physician
  * Optional biopsy approximately 14 days following initiation of neoadjuvant therapy
  Interventions: Procedure: Optional biopsy
- Cohort 2:Neoadjuvant endocrine + mammaglobin-A DNA vaccine (Experimental): * Will be treated with standard of care adjuvant endocrine therapy
  * Optional biopsy approximately 14 days following initiation of neoadjuvant therapy
  * Treated with 4 mg of mammaglobin-A DNA vaccine at 3 time points (Days 28, 56, and 84)
  * All study injections will be administered using a TriGrid electroporation device
  Interventions: Biological: Mammaglobin-A DNA Vaccine; Procedure: Optional biopsy
- Cohort 3: Neoadjuvant chemotherapy alone (Active Comparator): * Will be treated with standard of care neoadjuvant chemotherapy as determined by their treating physician
  * If archival tissue not sufficient, a research biopsy to obtain primary tissue must be done prior to day 28
  * Subjects who begin neoadjuvant endocrine therapy but are determined to not be responding at the Day 14 biopsy may begin chemotherapy treatment, at the discretion of the treating physician. These subjects may be enrolled in cohort 3
  Interventions: Procedure: Optional biopsy
- Cohort 4: Neoadjuvant chemotherapy + mammoglobin-A DNA vaccine (Experimental): * Will be treated with standard of care neoadjuvant chemotherapy as determined by their treating physician
  * If archival tissue not sufficient, a research biopsy to obtain primary tissue must be done prior to day 28
  * Treated with 4 mg of mammaglobin-A DNA vaccine at 3 time points (Days 28, 56, and 84)
  * All study injections will be administered using a TriGrid electroporation device
  * Subjects who begin neoadjuvant endocrine therapy but are determined to not be responding at the Day 14 biopsy may begin chemotherapy treatment, at the discretion of the treating physician. These subjects may be enrolled in either cohort 4
  Interventions: Biological: Mammaglobin-A DNA Vaccine; Procedure: Optional biopsy

INTERVENTIONS:
Biological: Mammaglobin-A DNA Vaccine
  Arms: Cohort 2:Neoadjuvant endocrine + mammaglobin-A DNA vaccine; Cohort 4: Neoadjuvant chemotherapy + mammoglobin-A DNA vaccine
Procedure: Optional biopsy

SUMMARY:
The purpose of this research study is to find out about the safety of injecting the gene (DNA) for mammaglobin-A into people with breast cancer. The DNA used in this study was purified from bacteria and contains the gene for mammaglobin-A. Mammaglobin-A is a protein that is highly expressed by breast cancer cells. Injection of mammaglobin-A DNA may be a way to generate an immune response to breast cancer cells. There is evidence that an immune response may be a way to fight cancer. In addition to evaluating the safety of the mammaglobin-A injection, this study is also looking at the immune response that the participant's body has after each injection.

ELIGIBILITY:
Inclusion Criteria:

A patient will be eligible for inclusion in this study only if ALL of the following criteria apply:

* Newly diagnosed histologically confirmed invasive breast cancer.
* Clinical T2-T4c, any N, M0 invasive ER+ (Allred Score of 6-8) and HER2- (0 or 1+ by IHC or FISH negative for amplification) breast cancer by AJCC 7th edition clinical staging, with the goal being surgery to completely excise the tumor in the breast and the lymph node. Patients with T1c tumors are eligible if they are considered candidates for neoadjuvant endocrine therapy or chemotherapy
* At least 1 measurable lesion.
* Candidate for neoadjuvant endocrine therapy or chemotherapy.
* At least 18 years of age.
* Eastern Cooperative Oncology Group (ECOG) performance status ≤2.
* Adequate organ and marrow function no more than 28 days prior to the start of neoadjuvant endocrine therapy or chemotherapy as defined below:

  * WBC ≥3,000/μL
  * absolute neutrophil count ≥1,500/μL
  * platelets ≥100,000/μL
  * total bilirubin ≤institutional upper limit of normal
  * AST/ALT ≤2.5 X institutional upper limit of normal
  * creatinine ≤ institutional upper limit of normal OR creatinine clearance ≥ 60 mL/min/1.73 m2 for patients with creatinine above IULN
* Postmenopausal or premenopausal. NOTE: Postmenopausal women, verified by: (1) bilateral surgical oophorectomy, or (2) no spontaneous menses ≥ 1 year or (3) no menses for <1 year with FSH and estradiol levels in postmenopausal range, according to institutional standards. Premenopausal women, verified by: (1) regular menses, or (2) FSH and estradiol levels in premenopausal range, according to institutional standards.
* Able to understand, and willing to sign a written informed consent document.
* Confirmation that primary tumor expresses mammaglobin-A by IHC.
* Clinical assessment by treating physician that the patient is responding to neoadjuvant therapy or umor Ki67 value is ≤ 10% after 14 days

Exclusion Criteria:

A patient will be ineligible for inclusion in this study if ANY of the following criteria apply:

* Received any of the following for treatment of this cancer (except for the neoadjuvant endocrine therapy or chemotherapy specified within this protocol):

  * Surgery
  * Radiation therapy
  * Chemotherapy
  * Biotherapy
  * Hormonal therapy
  * Investigational agent Note that subjects who do not respond initially to endocrine therapy may receive chemotherapy and remain on study.
* Receiving any other investigational agent(s) or has received an investigational agent within the last 30 days.
* Known metastatic disease.
* Known allergy, or history of serious adverse reaction to vaccines such as anaphylaxis, hives, or respiratory difficulty.
* Prior axillary lymph node sampling (sentinel lymph node biopsy or axillary lymph node dissection). FNA or core needle biopsy of axillary lymph node is acceptable.
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situation that would limit compliance with study requirements.
* Prior or currently active autoimmune disease requiring management with immunosuppression. This includes inflammatory bowel disease, ulcerative colitis, Crohn's disease, systemic vasculitis, scleroderma, psoriasis, multiple sclerosis, hemolytic anemia, immune-mediated thrombocytopenia, rheumatoid arthritis, systemic lupus erythematosus, Sjogren's syndrome, sarcoidosis, or other rheumatologic disease or any other medical condition or use of medication (e.g., corticosteroids) which might make it difficult for the patient to complete the full course of treatments or to generate an immune response to vaccines. Asthma or chronic obstructive pulmonary disease that does not require daily systemic corticosteroids is acceptable. Any patients receiving steroids should be discussed with the PI to determine if eligible.
* Pregnant or breastfeeding. A negative serum or pregnancy test is required no more than 7 days before study entry, and patients must be willing to employ adequate contraception. Women of childbearing potential must use two forms of contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation.
* Known HIV-positive status. These patients are ineligible because of the potential inability to generate an immune response to vaccines.
* Subjects with a strong likelihood of non-adherence such as difficulties in adhering to follow-up schedule due to geographic distance from the Siteman Cancer Center should not knowingly be registered.
* Individuals in whom a skinfold measurement of the cutaneous and subcutaneous tissue for the eligible injection sites (left and right medial deltoid region) exceeds 40 mm
* Individuals in whom the ability to observe possible local reactions at the eligible injection sites (deltoid region) is, in the opinion of the investigator, unacceptably obscured due to a physical condition or permanent body art
* Therapeutic or traumatic metal implant in the skin or muscle of either deltoid region.
* Acute or chronic, clinically significant hematologic, pulmonary, cardiovascular, or hepatic or renal functional abnormality as determined by the investigator based on medical history, physical examination, EKG, and/or laboratory screening test
* Any chronic or active neurologic disorder, including seizures and epilepsy, excluding a single febrile seizure as a child
* Syncopal episode within 12 months of screening
* Current use of any electronic stimulation device, such as cardiac demand pacemakers, automatic implantable cardiac defibrillator, nerve stimulators, or deep brain stimulators.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2015-01-07 (Actual); Primary Completion 2022-04-06 (Actual); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
Safety as measured by the number of participants who experience an adverse event | Day 126 (+/- 7days)
  Assessment of plasmid DNA safety will include both clinical observation and laboratory evaluation. Safety will be closely monitored after injection with eight or more clinical and laboratory assessments in the first 24 weeks of the trial. The following parameters will be assessed following vaccination:
  1. Local signs and symptoms
  2. Systemic signs and symptoms
  3. Laboratory evaluations, including blood counts and serum chemistries
  4. Adverse and serious adverse events
  Toxicity will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events v4.0

SECONDARY OUTCOMES:
Immune response | Week 52
  ELISPOT analyses and intracellular cytokine expression analyses using multi-parameter flow cytometry, and peptide MHC tetramer analyses will be performed. Peripheral blood will be obtained at two independent time points before vaccination (Pre-study, and Day 28 +/- 7 days), and at four independent time points following vaccination (Day 56 +/- 7 days, Day 84 +/- 7 days, Day 112 +/- 7 days, and Day 365 +/- 28 days).
Progression-free survival (PFS) | 5 years
  ◦Progressive disease - At least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study, appearance of one more new lesions PFS is defined as the duration of time from start of treatment to time of progression or death, whichever occurs first.
Overall survival (OS) | 5 years

OTHER OUTCOMES:
Objective tumor response rate (ORR) | 5 years
  -ORR=complete response (CR) + partial response (PR)
  * Complete response: disappearance of all lesions and normalization of tumor marker level
  * Partial response: at least a 30% decrease in the sum of the diameters of target lesions and no new lesions

CONTACTS AND LOCATIONS:
Overall Officials: William Gillanders, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu